CLINICAL TRIAL: NCT02525237
Title: Apatinib in Combination With S-1 as First-Line Treatment in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Apatinib in Combination With S-1 as First-Line Treatment in Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingdao Municipal Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaochun Zhang, Chairman, Qingdao Municipal Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-G316
Record Dates: First submitted 2015-08-11; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; S 1 (combination)

ARMS (1):
- Apatinib plus S-1 (Experimental): Apatinib (500 mg qd p.o.) concomitantly with S-1 (40 mg/m2 qd days 1-14 q3w p.o.)
  Interventions: Drug: Apatinib; Drug: S-1

INTERVENTIONS:
Drug: Apatinib — Apatinib (500 mg qd p.o.) until disease progression or intolerable toxicity
  Other Names: ATAN
Drug: S-1 — S-1 (40 mg/m2 qd days 1-14 q3w p.o.) until disease progression or intolerable toxicity

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Apatinib combined with S-1 as first-line therapy for patients with advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, aged ≥18 years;
2. Histologically confirmed adenocarcinoma of the stomach with inoperable locally advanced or recurrent and/or metastatic disease;
3. Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1);
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 3;
5. No previous chemotherapy for advanced/metastatic disease 1) Prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study); 2) No previous targeted therapy; 3) For patients who can't tolerate first-line chemotherapy or refuse to accept chemotherapy, if they request to participate in this study, may receive apatinib monotherapy after consultation with the principal investigator in consideration of ethics.
6. Hematological, Biochemical and Organ Functions: HB ≥ 80 g/L, ANC ≥ 1.5×109/L, PLT ≥ 80×109/L, BIL < 1.5×ULN, ALT or AST < 2.5×ULN (or < 5×ULN in patients with liver metastases), Serum Cr ≤ 1×ULN, Cr clearance ≥ 50 mL/min;
7. Life expectancy of more than 3 months;
8. Duration from operation is more than 4 weeks;
9. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.
10. Signed informed consent.

Exclusion Criteria:

1. Patients with poor-controlled arterial hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease, arrhythmia (including QT interval prolongation, for man > 450 ms, for woman > 470 ms), and cardiac dysfunction greater than Class II;
2. Factors affecting the oral medication, such as inability to swallow, chronic diarrhea and intestinal obstruction;
3. Patients with a clear tendency of gastrointestinal bleeding;
4. Abnormal coagulation function (INR > 1.5×ULN, APTT > 1.5×ULN), with tendency of bleed;
5. Pregnant or lactating women;
6. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Event driven, an expected average of 8 months
Safety will be assessed by incidence of adverse events | An expected average of 8 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | An expected average of 8 months
Disease control rate (DCR) | An expected average of 8 months
Overall survival (OS) | Event driven, an expected average of 24 months
Quality of life (QoL) | An expected average of 24 months
  Quality of life of patient will be measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 [EORTC QLQ-C30].